CLINICAL TRIAL: NCT04924686
Title: A Bacterial Bi-functional Peptidoglycan Hydrolase Sheds NOD2 Ligands to Regulate Gut Homeostasis
Brief Title: Changes of Muramyl Dipeptide in Intestinal and Extra-intestinal Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Hongwei Zhou, Proffessor, Zhujiang Hospital
Other Study IDs: ZhujiangH-1
Record Dates: First submitted 2021-06-07; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Cancer; Inflammatory Bowel Disease; Atherosclerotic Cardiovascular Disease; Type2 Diabetes Mellitus
Keywords: NOD2 ligands
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fecal, Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Crohn's disease: The fecal and plasma were collected
  Interventions: Other: Observational studies, no intervention
- Ulcerative colitis: The fecal and plasma were collected
  Interventions: Other: Observational studies, no intervention
- Diabetes mellitus, type 2: The fecal and plasma were collected
  Interventions: Other: Observational studies, no intervention
- Atherosclerotic cardiovascular disease: The fecal and plasma were collected
  Interventions: Other: Observational studies, no intervention
- Colorectal cancer: The fecal and plasma were collected
  Interventions: Other: Observational studies, no intervention

INTERVENTIONS:
Other: Observational studies, no intervention — Observational studies, no intervention

SUMMARY:
Nucleotide-binding oligomerization domain 2 (Nod2) signaling is critical for human health.To figure out the clinical relevance of NOD2 ligands, the investigators plan to evaluate the change of NOD2 ligands in inflammatory bowel diseases (IBD), CRC, atherosclerotic cardiovascular disease (ACVD), and type 2 diabetes mellitus (DM2 ).

DETAILED DESCRIPTION:
Previous studies have shown that NOD2 gene mutants were associated with the Crohn's disease (CD), colorectal cancer (CRC) and many other diseases, suggesting the critical role of NOD2 signaling in human physiology and pathogenethesis. However, whether decreased NOD2 ligands also contributed to these diseases is unknown. In this study, the investigators plan to evaluate the change of NOD2 ligands in inflammatory bowel diseases (IBD), CRC, atherosclerotic cardiovascular disease (ACVD), and type 2 diabetes mellitus (DM2 ). For each of the patient, a sex- and age- matched control were chosen. Both the targeted metabolomics (LC-MS-MS methods) and NOD2-transfected cells co-expressing NF-κB luciferase reporters were used to test NOD2 ligands in the fecal and plasma samples.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females at least 18-70 years old.
2. Patient able to give informed consent.
3. Patient with biopsy-proven CRC
4. Patient with biopsy-proven Crohn's disease (CD) or ulcerative colitis(UC), in the active phase.
5. patients with clinical diagnosed DM2
6. patients with ACVD:coronary angiography more than 50% stenosis in single or multiple vessels.
7. The age- and sex- matched health controls for each patient.

Exclusion Criteria:

1.Use antibiotics or probiotics within the last 2 weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the patients with IBD, CRC, ACVD or DM2 hospitalized in Zhujiang hospital will be eligible to be enrolled. Also, their age- and sex- matched healthy controls making a physical examination in Zhujiang hospital will be eligible to be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-05-10 (Actual); Primary Completion 2023-06-10 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
NOD2 ligands in fecal and plasma | baseline
  detected using targeted metabolomics (LC-MS-MS methods) and NOD2-transfected cells co-expressing NF-κB luciferase reporters

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhou, professor, Principal Investigator — Zhujiang Hospital, Guangzhou, Guangdong
Locations (1):
- Zhujiang hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Philpott DJ, Sorbara MT, Robertson SJ, Croitoru K, Girardin SE. NOD proteins: regulators of inflammation in health and disease. Nat Rev Immunol. 2014 Jan;14(1):9-23. doi: 10.1038/nri3565. Epub 2013 Dec 13. PMID 24336102